CLINICAL TRIAL: NCT04192565
Title: Endoscopic Resection of Colorectal Lesions with ColubrisMX Endoluminal Surgical System (ELS for Its Initials in English), Prospective Clinical Study
Brief Title: A Prospective Investigation of the ColubrisMX ELS System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ColubrisMX (Industry)
Collaborators: Faculdade de Medicina do ABC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMX-CSP-CS002
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Neoplasms; Colorectal Polyp; Colorectal Adenoma; Colorectal Adenomatous Polyp
Keywords: Colorectal Neoplasms; Colorectal Polyp; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Robotic Transanal Endoluminal Resection (Experimental): Robotic Transanal Endoluminal Resection of Colorectal Lesions
  Interventions: Device: ColubrisMX Endoluminal Surgical (ELS) System

INTERVENTIONS:
Device: ColubrisMX Endoluminal Surgical (ELS) System — Robotic Transanal Endoluminal Resection of Colorectal Lesions using the ColubrisMX Endoluminal Surgical (ELS) System

SUMMARY:
This study is a prospective, single-arm, open-label, multi-center, feasibility study to evaluate the safety and efficacy of the ColubrisMX ELS System in patients undergoing transanal endoluminal procedures, specifically colorectal Endoscopic Submucosal Dissection.

DETAILED DESCRIPTION:
Endoscopic resection of small polyps is performed routinely through conventional outpatient colonoscopy. Larger polyps or incipient tumors can be excised with endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD). These minimally invasive procedures have been shown to be viable alternatives to conventional surgical resections with less risk of complications, shorter hospital stay and lower costs.

Both flexible endoscopic and open/laparoscopic surgical approaches have procedural limitations that can have considerable impact on patient care. Traditional endoscopic tools have technical inadequacies that may inhibit the physician's ability to complete more complex tasks consistent with a surgical technique. Conversely, a traditional open or laparoscopic surgical approach involves increased risk of complications (such as surgical site infection), increased pain and blood loss, longer recovery, and surgical scars. The objective of this clinical study is to assess the safety and efficacy of the ColubrisMX Endoluminal Surgical (ELS) System, a new robotic technology designed to assist the physician with precision, flexibility, and control during endoluminal removal of colorectal lesions.

ELIGIBILITY:
INCLUSION CRITERIA

All of the following criteria must be present to be eligible for the study:

1. Aged 18-75 years
2. BMI ≤ 35 kg/m2
3. Patient agrees to participate in the study by giving signed informed consent
4. Benign lesions of the rectum, such as adenoma, submucosal nodule, or polyp
5. Mucosal neoplasm
6. Eligible to undergo standard endoscopic submucosal dissection.
7. Patient reviewed and approved by Local Oncology Committee to undergo robotic procedure.

EXCLUSION CRITERIA

Patients will be excluded from the study if any of the following criteria are present:

Preoperative

1. Anatomy unsuitable for endoscopic visualization or endoluminal surgery
2. Extensive previous surgery in the lower GI tract
3. Prior radiation treatment for colorectal cancer
4. Patient with distant metastases
5. Untreated active infection
6. Vulnerable population (e.g., prisoners, mentally disabled)
7. Severe concomitant illness (i.e., cancer) that drastically shortens life expectancy or increases risk of therapeutic interventions
8. Breastfeeding or pregnant, or intend to become pregnant during the course of the study
9. Currently enrolled in or discontinued within the last 30 days from a clinical trial of an investigational drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
10. In the opinion of the Investigator, the patient is unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
11. Patients with immunosuppression drugs (chemotherapy) due to an increase potential infection and poor healing
12. Patients with a high cardiac or pulmonary risk (these patients require clearance from a cardiologist and pulmonologist)
13. Preoperative blood thinner i.e., coumadin or heparin.
14. Obstructing rectal cancer
15. History of inflammatory bowel disease

Intraoperative

1. Existing stricture or anatomical blockage in lower GI tract preventing overtube from reaching desired position.
2. Disease is more extensive and not amenable to standard ESD
3. Inadequate bowel prep
4. Complex anatomical findings not feasible for endoscopic approach

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-13 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of success (%) | 24 hours post-op
  Percentage of patients with no conversion during surgery and no major complications (Clavien-Dindo ≥ III complication rating) for 24 hours post-op.
Rate of conversions (%) | Intraoperative
  Percentage of patients with a change in treatment plan to a conventional open or laparoscopic procedure.
Estimated blood loss (mL) | Intraoperative
  Estimated amount of intraoperative blood loss (up to the point of needing transfusion).
Operative time (min) | Intraoperative
  Duration from transanal insertion of the robotic flexible overtube to final removal of the flexible overtube from the anal verge.
Patients requiring transfusion (%) | Intraoperative
  Percentage of patients requiring transfusion during surgery.
Complication rate (%) | 60 Days
  Percentage of patients having Clavien-Dindo ≥ III intraoperatively or postoperatively at Days 7, 30, or 60.
Readmission rate (%) | 60 Days
  Percentage of patients with readmission that can be linked to colorectal submucosal dissection.
Major Adverse Events (MAE) during the first 60 days | 60 Days
  Freedom from procedural-related MAE, defined as a combined clinical endpoint of death or reoperation for failed surgical repair.

OTHER OUTCOMES:
En bloc resection rate (%) | Intraoperative
  Percentage of samples dissected en bloc, as assessed by the pathologist during postoperative assessment.
Rate of positive surgical lateral margins (PSLM) (%) | 60 Days
  The number and percentage of subjects with PSLM will be presented separately by subjects undergoing rectal ESD.
Rate of perforations repaired operatively (%) | Intraoperative
  Rate of perforations requiring repair through open or laparoscopic surgery.
Rate of perforations requiring repair through open or laparoscopic surgery (%) | Intraoperative
  Rate of perforations requiring repair through open or laparoscopic surgery
Rate of delayed perforations (%) | 60 Days
  Perforations that present 10 to 24 hours after procedure with clinical signs and symptoms of peritonitis.
Adverse Events | 60 Days
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in patients, users, or other persons, whether related to the investigational medical device.
Vital Signs | 60 Days
  Changes in vital signs from baseline to post-operative Days 7, 30 and 60.
Laboratory Assessments | 60 Days
  Changes in laboratory parameters and normal/abnormal status changes in laboratory parameters from baseline to post-operative Days 7, 30 and 60.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Grecco, MD, Principal Investigator — Faculdade de Medicina do ABC
Locations (1):
- Faculdade de Medicina do ABC, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No